CLINICAL TRIAL: NCT04016922
Title: Effect of Maternal Iron Deficiency Anemia on Fetal Hemodynamics and Neonatal Outcome
Brief Title: The Effect of Maternal Iron Deficiency Anemia on Fetal Hemodynamic and Neonatal Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Amin, Assistant lecturer, Cairo University
Other Study IDs: Fetal hemodynamics, neonates
Record Dates: First submitted 2019-06-24; First posted 2019-07-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Fetal Conditions
Keywords: Fetal hemodynamics.; Intrauterine growth restriction; Amniotic fluid index
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients with mild anemia (Hb concentration: 9.0-10.9 g\dl).
  Interventions: Other: Oral ferrous fumerate for Group A, Parenteral iron sucrose for Group B, Compatible blood transfusion for Group C
- Group B: Patients with moderate anemia (Hb concentration: 7.0-8.9 g\dl).
  Interventions: Other: Oral ferrous fumerate for Group A, Parenteral iron sucrose for Group B, Compatible blood transfusion for Group C
- Group C: Patients with severe anemia (Hb concentration: >7.0 g\dl).
  Interventions: Other: Oral ferrous fumerate for Group A, Parenteral iron sucrose for Group B, Compatible blood transfusion for Group C

INTERVENTIONS:
Other: Oral ferrous fumerate for Group A, Parenteral iron sucrose for Group B, Compatible blood transfusion for Group C — Consent, history. US: fetal heart activity, placental site, fetal biometry, AFI, anomalies, Doppler: umbilical artery, MCA, fetal renal artery, C\U ratio.
  * Maternal Hb,US at time of first visit, 10 days later after initiation of treatment, at EDD .
  * As part of routine medical care of these patients, they are managed as:
  A: give oral iron in the form of ferrous fumerate with the possible side effects. if Hb returns to normal, continue iron for 3 mon.
  B: admit to receive IV iron sucrose according to product literature allergic reaction may happen; antiallergic measures. C: give blood transfusion in the form of packed RBC. allergic and pyrogenic reaction and infection may occur. At delivery will be subjected to: examination, investigations, US.
  Other Names: routine medical care

SUMMARY:
This study will be conducted to show the effect of different degrees of maternal iron deficiency anemia on fetal hemodynamics and neonatal outcome and to evaluate the effect of treatment.

DETAILED DESCRIPTION:
Hemoglobin concentration is used to determine the diagnosis and severity of anemia in low resource settings, an indicator that is routinely screened using WHO-defined hemoglobin cutoffs. These thresholds are lower for pregnant women (females ≥ 15 years of age) than non-pregnant women (11.0 g/dl versus 12.0 g/dl). Severity of anemia is determined using additional cutoffs, with severe anemia defined as a hemoglobin level of less than 7.0 g/dl.

Iron deficiency is defined as a condition in which there are no mobilizable iron stores, resulting from a long-term negative iron balance and leading to a compromised supply of iron to the tissues. Finally, the most significant negative consequence of ID is anemia, usually microcytic hypochromic in nature.

IDA has been linked to unfavorable outcomes of pregnancy. It is the most common nutritional disorder in the world affecting two billion people worldwide with pregnant women particularly at risk. According to WHO report, 2001 indicates that IDA is a significant problem throughout the world ranging from 35-75% in developing countries (average 56%) whereas in industrialized countries the average prevalence is 14%.

Distribution of blood flow (between the placental and cerebral regions) is determined with Middle cerebral artery PI/Umbilical artery PI (C/U ratio); this parameter is always > 1.1 during normal pregnancy, but decreases in the case of hypoxia because of umbilical artery resistance index increase (increase in placental resistance) and cerebral resistance index decrease (cerebral vasodilation).

Perinatal morbidity & mortality of IUGR infants is 3-20 times greater than normal infants. These cases may be followed with outpatient monitoring and they often deliver at term. However process is not severe enough to stop fetal growth completely or to deteriorate. The umbilical artery and the middle cerebral artery waveforms may be abnormal, without effect is seen on Doppler and growth until 26-32 weeks gestation; Mild utero-placental insufficiency.

Iron deficiency and iron deficiency anemia during pregnancy are risk factors for preterm delivery, prematurity and small for gestational age birth weight. Iron deficiency has a negative effect on intelligence and behavioral development in the infant. It is essential to prevent iron deficiency in the fetus by preventing iron deficiency in the pregnant woman.

Prevention and control is typically achieved through iron fortification of food staples like flour and rice and/or through administration of iron supplements most often in iron tablets. Although iron supplements are widely available and fortified foods constitute a major component of the diet in the developed world, access is limited in the developing world

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females aged 20- 35 years.
* Gestational age 32 weeks or more.
* Living singleton fetus.

Exclusion Criteria:

* Multifetal pregnancy.
* Patients with chronic illness or medical disorders other than iron deficiency anemia.
* Patients with history of recurrent perinatal deaths or recent blood transfusion or other vitamin deficiency anemia.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: * The pregnant women were divided into three groups:
  1. Group A : Patients with mild anemia (Hb concentration: 9.0-10.9 g\dl).
  2. Group B : Patients with moderate anemia (Hb concentration: 7.0-8.9 g\dl).
  3. Group C : Patients with severe anemia (Hb concentration: >7.0 g\dl).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Changes in fetal vascular doppler parameters. | 4 months from June 2019 till October 2019
  Fetal doppler parameters by resistance index and pulsatility index at first visit and 10 days after recieving treatment and at delivery.
Neonatal birth weight | 4 months June 2019 till October 2019
  Neonatal birth weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Muhamad Ehab, professor, Study Chair — Cairo University
Locations (1):
- Kasralainy hospital, Giza, Egypt

REFERENCES:
- [Background] Breymann C. Iron Deficiency Anemia in Pregnancy. Semin Hematol. 2015 Oct;52(4):339-47. doi: 10.1053/j.seminhematol.2015.07.003. Epub 2015 Jul 10. PMID 26404445
- [Background] Abu-Ouf NM, Jan MM. The impact of maternal iron deficiency and iron deficiency anemia on child's health. Saudi Med J. 2015 Feb;36(2):146-9. doi: 10.15537/smj.2015.2.10289. PMID 25719576
- [Background] Breymann C; Anaemia Working Group. [Current aspects of diagnosis and therapy of iron deficiency anemia in pregnancy]. Praxis (Bern 1994). 2001 Aug 2;90(31-32):1283-91. German. PMID 11519193
- [Background] Lee AI, Okam MM. Anemia in pregnancy. Hematol Oncol Clin North Am. 2011 Apr;25(2):241-59, vii. doi: 10.1016/j.hoc.2011.02.001. PMID 21444028
- [Background] Rasmussen K. Is There a Causal Relationship between Iron Deficiency or Iron-Deficiency Anemia and Weight at Birth, Length of Gestation and Perinatal Mortality? J Nutr. 2001 Feb;131(2S-2):590S-601S; discussion 601S-603S. doi: 10.1093/jn/131.2.590S. PMID 11160592